CLINICAL TRIAL: NCT05924165
Title: Narcotic-Free Percutaneous Nephrolithotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mantu Gupta, Professor of Urology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-23-00206
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis | interventions — Oxycodone; Ketorolac

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Operating surgeon will be blinded to treatment arm intraoperatively (will not be blinded postoperatively)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid group (Active Comparator): Patients will be prescribed 5mg Oxycodone, Q6 PRN postoperatively.
  Interventions: Drug: 5mg Oxycodone, Q6 PRN
- NSAID (Active Comparator): Patients will be prescribed 10mg Ketorolac, Q6 PRN postoperatively.
  Interventions: Drug: 10mg Ketorolac, Q6 PRN

INTERVENTIONS:
Drug: 5mg Oxycodone, Q6 PRN — Oxycodone is an opioid that is used to relieve moderate to severe pain.
  Arms: Opioid group
Drug: 10mg Ketorolac, Q6 PRN — Ketorolac is an NSAID used to relieve moderately severe pain.
  Arms: NSAID

SUMMARY:
This is a randomized control trial comparing oral ketorolac and opioid medication for the use of post-operative analgesia.

DETAILED DESCRIPTION:
This is a randomized control trial comparing oral ketorolac (10mg, Q6 PRN) and oxycodone (5mg, Q6 PRN) medication for the use of post-operative analgesia after kidney stone removal surgery called percutaneous nephrolithotomy (PCNL). Primary endpoints are visual analog pain scores (VAS) for days 1-5 and day 10 post operatively. Secondary endpoints are pill counts, patient-related outcome survey (PROMIS) scores, emergency room visits, and patient telephone calls. 90 subjects will be enrolled, with 45 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing scheduled unilateral standard (24Fr), PCNL with at least 2cm stone burden, with expected single access

Exclusion Criteria:

* Pregnant women
* History of chronic opioid abuse
* Allergy, hypersensitivity, or other contraindication to NSAID usage such as

  * eGFR < 60 mL/min
  * Peptic ulcer disease or history of gastric bypass
  * Concurrent use of antiplatelet or anticoagulation therapy (including aspirin)
  * Thrombocytopenia
  * Suspected or confirmed cerebrovascular bleeding, patients with hemorrhagic diathesis, incomplete hemostasis, and those at high risk of bleeding.
  * Concomitant medications:

    * Other NSAIDs
    * Antiplatelet or anticoagulation medications
    * Probenecid
    * Pentoxifylline
* Allergy, hypersensitivity, or other contraindication to opioids:

  * Current opioid prescription/usage for any reason, including active treatment with suboxone or methadone
  * Respiratory depression
  * Patients with acute or severe bronchial asthma or hypercarbia
  * Patients who have or is suspected of having paralytic ileus as PCNL done under general anesthesia
  * Patients with hepatic Impairment
  * Concomitant medications:

    * Monoamine Oxidase Inhibitors (MAOIs)
    * Mixed Agonist/Antagonist and Partial Agonist Opioid Analgesics
* Diagnosis of chronic pain disorder
* Reduced sensation of abdomen or pelvis (e.g. patients with spinal cord injury)
* Pre-existing stent or nephrostomy tube
* Urinary tract anomalies such as urinary diversion, horseshoe kidney, solitary kidney, urinary stricture disease, ureteropelvic junction obstruction, pelvic kidney, stone in calyceal diverticulum)
* Pulmonary disease
* Liver disease
* Seizure disorders
* Subjects taking nephrotoxic medications
* Subjects taking medications that can increase sedation risk (benzodiazepines or other sedative hypnotics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mantu Gupta, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from 5-19-2023 to 12-26-2024
Groups:
- Opioid Group: Patients prescribed 5mg Oxycodone, Q6 as needed (PRN) postoperatively.
  5mg Oxycodone, Q6 PRN: Oxycodone is an opioid that is used to relieve moderate to severe pain.
- NSAID: Patients prescribed 10mg Ketorolac, Q6 PRN postoperatively.
  10mg Ketorolac, Q6 PRN: Ketorolac is an NSAID used to relieve moderately severe pain.
Period: Overall Study
Arm/Group | Opioid Group | NSAID
Started | 45 | 45
Completed | 43 | 42
Not Completed | 2 | 3
Not completed — Physician Decision | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Opioid Group: Patients prescribed 5mg Oxycodone, Q6 PRN postoperatively.
  5mg Oxycodone, Q6 PRN: Oxycodone is an opioid that is used to relieve moderate to severe pain.
- Total: Total of all reporting groups
Arm/Group | Opioid Group | NSAID | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [57 to 70] | 63 [45 to 74] | 64 [51 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 25 | 24 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 32 | 32 | 64
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 26 | 25 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 20
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 27.98 [24.14 to 31.38] | 27.42 [25.07 to 31.94] | 27.46 [25.02 to 31.76]

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Pain Scores
Description: Visual Analog Scale (VAS) to measure pain: The minimum score of '0' indicates "no pain" and the maximum score of '10' indicates "Worst pain imaginable" along a line. Participants will be asked to mark the level of their pain along the line. Visual analog scale (VAS) pain scores will be recorded
Time Frame: post-op day 5 and post-op day 10
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Opioid Group | NSAID
Number analyzed (Participants) | 43 | 42
score on a scale
  post-op day 5 | 4.5 [3 to 7] | 5 [3 to 6]
  post-op day 10 | 1 [0 to 2] | 1 [0 to 3]

2. Secondary Outcome: Pill Count
Description: A pill count will be conducted of each prescribed postoperative medication.
Time Frame: post-op at day 10
Measure: Mean (Standard Deviation); unit: pills
Arm/Group | Opioid Group | NSAID
Number analyzed (Participants) | 43 | 42
pills | 6.5 (5) | 12 (6)

3. Secondary Outcome: Number of Participants Who Called the Office
Description: Number of participants with pain related calls to the office recorded.
Time Frame: post-op up to day 10
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Group | NSAID
Number analyzed (Participants) | 43 | 42
Participants | 5 | 8

4. Secondary Outcome: Number of Participants With Pain Related Visits
Description: Number of participants with pain related visits to the office or Emergency Department (ED) visits recorded.
Time Frame: post-op up to day 10
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Group | NSAID
Number analyzed (Participants) | 43 | 42
Participants | 3 | 2

5. Secondary Outcome: Patient-related Outcome Survey (PROMIS) Scores
Description: Patients given a survey containing questions from Patient-related outcome survey (PROMIS) instruments.
  A series of person-centered measures that evaluate and monitor physical, mental, and social health in adults and children. 10-item patient-reported questionnaire. standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
Time Frame: post-op at day 10
Measure: Median (Inter-Quartile Range); unit: T-score
Arm/Group | Opioid Group | NSAID
Number analyzed (Participants) | 43 | 42
T-score | 10 [7 to 13] | 10 [8 to 15]

ADVERSE EVENTS:
Time Frame: up to 10 days post-op
Description: There were no adverse events.
Arm/Group | Opioid Group | NSAID
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT05924165/Prot_SAP_001.pdf
  • Informed Consent Form (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT05924165/ICF_000.pdf